CLINICAL TRIAL: NCT05131776
Title: Concurrent EUS-guided Intra-tumour Injection of OncoSil (32P) With Chemotherapy in Locally Advanced Pancreatic Carcinoma.
Brief Title: EUS-guided Intra-tumour Injection of OncoSil for Locally Advanced Pancreatic Carcinoma.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTEC-2021-0234
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer; Endoscopic Ultrasound
Keywords: Pancreatic cancer; Endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: OncoSil™ is comprised of OncoSil Phosphorous-32 Microparticles (hereafter Microparticles) and OncoSil Diluent (hereafter Diluent). OncoSil™ is an active implantable (radiological) medical device intended for use in brachytherapy, where cancer is treated by the insertion of radioactive implants directly into the cancerous tissue. OncoSil™ has been designed to be injected directly into, and to deliver an average absorbed dose of 100 Gy to the target treatment tumour. In therapeutic use 98% of the radiation is delivered within 81 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EUS-guided oncosil injection (Experimental): All patients will receive OncoSilTM during the 4th week of the first chemotherapy cycle.
  Interventions: Device: EUS-guided oncosil injection

INTERVENTIONS:
Device: EUS-guided oncosil injection — All patients will receive OncoSilTM during the 4th week of the first chemotherapy cycle.

SUMMARY:
The outcomes of concurrent EUS-guided intra-tumour injection of P-32 microparticles (OncoSil; OncoSil Medical, Australia) with chemotherapy in locally advanced pancreatic carcinoma in the local population is uncertain.

The aim of the current study is to assess efficacy and safety of the intervention in the local population. We hypothesis that the intervention is safe and useful for tumour downstaging.

DETAILED DESCRIPTION:
This would be a cohort study including patients with locally advanced pancreatic cancer medically fit to receive chemotherapy. Eligible patients would receive gemcitabine (GNP; 28- day cycles). P-32 microparticles (OncoSil; OncoSil Medical) implantation will be planned at weeks 4-5. P-32 activity will be calculated from patients' tumor volume (TV) to deliver 100 Gy absorbed dose, with implantation assessment by EUS and Bremsstrahlung SPECT/CT imaging. The primary endpoint was safety and tolerability, graded using CTCAE v4.0. Response will be assessed using RECIST 1.1 with 8-weekly CT scans and FDG-PET scans at baseline and week 12. The outcome parameters include adverse events, response of the tumour, local progression free survival and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Study participants are ≥ 18 years of age at screening.
2. Histologically or cytologically proven adenocarcinoma of the pancreas.
3. Unresectable locally advanced pancreatic carcinoma. Patients with technically resectable tumours (T1-T3) will also be eligible, if they are deemed unresectable due to medical comorbidities or refusal of surgery.
4. Pancreatic target tumour diameter ≥ 2.0 cm (shortest axis) to ≤ 6.0 cm (longest axis)
5. An ECOG Performance Status of 0 to 1 and Karnofsky Performance Status of 80 - 100.
6. Willing and able to complete study procedures within the study timelines.
7. Adequate renal function: serum creatinine less than 1.5 x upper limit of normal (ULN).
8. Adequate liver function: Serum SGOT/AST and serum SGPT/SLT < 3 times ULN and serum bilirubin <1.5 times the ULN unless the patient is known to have prior Gilbert's Syndrome.
9. Adequate bone marrow function: white blood cells (WBCs) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, haemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/mm3.
10. Life expectancy of at least 3 months at the time of screening as judged by the investigator.
11. Not pregnant, and if of childbearing potential, agrees to use adequate birth control (hormonal or barrier method of birth control or abstinence) prior to study entry and during the study and agrees not to donate sperm or ova, for the duration of the study and 12 months post implantation of the investigational device.
12. Provide signed Informed Consent.
13. Technically feasible - tumour must be within reach of the EUS probe for fine needle Injection.

Exclusion Criteria:

1. More than one primary lesion.
2. Any prior radiotherapy or chemotherapy for pancreatic cancer.
3. Use of other investigational agent at the time of screening, or within 30 days or five half-lives of Screening Visit 1, whichever is longer.
4. History of malignancy, treated or untreated, within the past five years whether or not there is evidence of local recurrence or metastases, with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ.
5. Evidence of tumour invasion into stomach, duodenum or peritoneum
6. In the opinion of the investigator, EUS directed implantation posing undue study participant risk. This includes:

   1. Where previous EUS-FNA was considered technically too difficult to perform;
   2. Imaging demonstrates multiple collateral vessels surrounding or adjacent to the target tumour within the pancreas;
   3. Presence (or significant risk) of varices near to the target tumour.
7. A known allergy or history of hypersensitivity to silicon, Phosphorus or any of the OncoSil™ components.
8. Patients who do not consent to chemotherapy
9. Actively on medication that increase bleeding risk (i.e. aspirin, clopidogrel, warfarin, NOAC).
10. Any other health condition that would preclude participation in the study in the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 30 day
  Any untoward medical occurrence, unintended disease or injury, oruntoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival of the patient
Local Disease Control Rate | 16 week
  proportion of study participants whose local tumour response is stable disease (SD), partial response (PR), or complete response (CR)
Local Progression Free Survival | 6 months
  the time from enrolment to the date of the radiological scan used to determine local tumour progression or date of death, whichever comes first.
Progression Free Survival | 5 years
  the time from enrolment to the date of tumour progression or of recurrence (in case of complete response (CR))

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Result] Rosemurgy A, Luzardo G, Cooper J, Bowers C, Zervos E, Bloomston M, Al-Saadi S, Carroll R, Chheda H, Carey L, Goldin S, Grundy S, Kudryk B, Zwiebel B, Black T, Briggs J, Chervenick P. 32P as an adjunct to standard therapy for locally advanced unresectable pancreatic cancer: a randomized trial. J Gastrointest Surg. 2008 Apr;12(4):682-8. doi: 10.1007/s11605-007-0430-6. Epub 2008 Feb 12. PMID 18266048